CLINICAL TRIAL: NCT05542355
Title: A Phase 1, Multicentre, 2-Part, Randomised, Parallel-arm, Placebo-controlled, Partially Double-blind Study to Evaluate the Safety and Target Engagement of EXL01 in the Maintenance of Steroid-induced Clinical Response or Remission in Participants With Mild to Moderate Crohn's Disease
Brief Title: EXL01 in the Maintenance of Steroid-induced Clinical Response/Remission in Participants With Mild to Moderate Crohn's Disease
Acronym: MAINTAIN
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to low recruitment
Sponsor: Exeliom Biosciences (Industry)
Collaborators: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EXL01-CD-001; 2021-003432-81 (EudraCT Number)
Record Dates: First submitted 2022-09-02; First posted 2022-09-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Crohn Disease
Keywords: Gastrointestinal Diseases; Inflammatory Bowel Disease; Colonic Diseases; Intestinal Diseases; Digestive System Diseases; Microbiota; Crohn Disease, remission; Faecalibacterium prausnitzii
MeSH Terms: conditions — Crohn Disease; Gastrointestinal Diseases; Inflammatory Bowel Diseases; Colonic Diseases; Intestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: Part A = Single Arm open label. Part B = Randomised, placebo-controlled, double-blind.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part A: None (Open-label). Part B: Double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (Open-Label EXL01 Maintenance Therapy) (Experimental): Oral EXL01 once daily for up to 24 weeks (after SoC corticosteroid induction therapy).
  Interventions: Drug: EXL01; Other: SoC corticosteroid - Induction Period; Other: SoC corticosteroid - Tapering
- Part B (EXL01 Maintenance Therapy) (Experimental): Oral EXL01 once daily for up to 24 weeks (after SoC corticosteroid induction therapy).
  Interventions: Drug: EXL01; Other: SoC corticosteroid - Induction Period; Other: SoC corticosteroid - Tapering
- Part B (Placebo Maintenance Therapy) (Placebo Comparator): Oral EXL01 matched placebo once daily for up to 24 weeks (after SoC corticosteroid induction therapy).
  Interventions: Drug: Placebo; Other: SoC corticosteroid - Induction Period; Other: SoC corticosteroid - Tapering

INTERVENTIONS:
Drug: EXL01 — Oral EXL01 once daily for up to 24 weeks (after SoC corticosteroid induction therapy).
  Other Names: Faecalibacterium prausnitzii EXL01-strain
  Arms: Part A (Open-Label EXL01 Maintenance Therapy); Part B (EXL01 Maintenance Therapy)
Drug: Placebo — Oral EXL01 matching placebo once daily for up to 24 weeks (after SoC corticosteroid induction therapy).
  Arms: Part B (Placebo Maintenance Therapy)
Other: SoC corticosteroid - Induction Period — Oral prednisone 40 mg or budesonide 9 mg once daily for 3 to 7 weeks, as assigned by the investigator
Other: SoC corticosteroid - Tapering — Same product as the Induction Period.
  Oral prednisone: 30 mg for 1 week, 25 mg for 1 week, 20 mg for 1 week, 15 mg for 1 week, 10 mg for 1 week, 5 mg for 1 week and stop.
  OR
  Oral budesonide: 6 mg for 3 weeks, 3 mg for 3 weeks, stop.

SUMMARY:
A Phase 1, 2-part, multicentre study to evaluate the safety and preliminary efficacy of the oral administration of EXL01 in the maintenance of corticosteroid-induced clinical response/remission in participants with mild to moderate Crohn's Disease (CD).

DETAILED DESCRIPTION:
Initially, all participants will received standard of care (SoC) corticosteroid induction therapy for 3 to 7 weeks. Participants who meet the protocol defined criteria for response after corticosteroid therapy will enter a Maintenance Period. Participants not in clinical response/remission at the end of the Induction Period will discontinue the study without further study treatment. In the Maintenance Period, participants will receive oral EXL01 or placebo in combination with corticosteroid treatment (that is progressively tapered) and be monitored for safety and efficacy.

The study will be conducted in 2 parts:

* Part A: Participants eligible for maintenance treatment will receive open-label oral EXL01 for up to 24 weeks.
* Part B: Participants eligible for maintenance treatment will be randomised 2:1 to receive double blind oral EXL01 or placebo for up to 24 weeks.

Participants will be monitored for 30 days after end-of-treatment.

Due to the low recruitment rate into Part A, the study was discontinued early; Part B did not start.

ELIGIBILITY:
Key Inclusion Criteria:

Must meet all of the following criteria at the start of the Induction Period:

* Male or female aged ≥18 years and <75 years at the time of providing informed consent.
* A diagnosis of CD with ileal involvement for at least 3 months prior to Screening.
* A CDAI score >180 and <350.
* Part B only: Active mucosal inflammation.

Key Exclusion Criteria:

* Stricture with obstructive syndrome <3 months prior to Screening.
* Stenosis making endoscopic access to the terminal ileum difficult.
* Received treatment with high dose corticosteroid (≥40 mg prednisone daily) for >5 weeks within 3 months prior to Screening.
* Part B only: Received >3 prior biologic treatments or JAK inhibitors for CD including infliximab, ustekinumab, vedolizumab, adalimumab, certolizumab, risankizumab, and upadacitinib.
* Major surgery or significant trauma ≤4 weeks prior to Screening.
* Small bowel resection >1 m in total or clinical manifestations of short bowel syndrome.
* Current stoma (ileostomy or a colostomy) or had a stoma in the last 6 months or any other intraabdominal surgery within 3 months prior to Screening.
* Started or stopped immunosuppressive therapy (thiopurine, methotrexate, tacrolimus, or other classical immunosuppressant) within 3 months prior to Screening.
* Received faecal microbial transplant within 3 months prior to Screening.
* Systemic infection or other serious infection requiring systemic treatment within 30 days prior to Screening.
* Pregnant, breastfeeding, or expecting to conceive during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
The systemic and intestinal safety and tolerability of orally administered EXL01 | Up to 43 weeks
  Number of participants with adverse events (AE[s]). Number of participants with treatment discontinuations due to an AE. AEs assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Proportion of participants in steroid-free clinical remission at Week 24 | Maintenance Period Week 24
  Endpoints: Crohn's disease activity index (CDAI) score (higher scores indicate more active/severe disease) and use of corticosteroids
Proportion of participants in steroid-free clinical remission and mucosal healing at Week 24 | Maintenance Period Week 24
  This is a composite measure. Endpoints: CDAI score, simple endoscopic score for Crohn's Disease (SES-CD; higher scores indicate more severe disease), and use of corticosteroids
Proportion of participants in steroid free clinical remission and mucosal healing and normal inflammatory markers at Week 24 | Maintenance Period Week 24
  This is a composite measure. Endpoints: CDAI score, SES-CD score, C-reactive protein (CRP) level (a marker of inflammation), faecal calprotectin level (a marker of intestinal inflammation), and use of corticosteroids
Proportion of participants with an endoscopic response at Week 24 | Maintenance Period Week 24
  Endpoint: SES-CD score
Time to clinical relapse in participants with CD treated with EXL01 to participants treated with placebo (Part B only) | Maintenance Period Baseline to Week 24
  Time to clinical relapse, defined as the time from first dose of EXL01 or placebo to first documented clinical relapse (Part B only)
Comparison of the SES-CD and histology of the intestinal mucosa in participants with CD treated with EXL01 to participants treated with placebo (Part B only) | Maintenance Period Baseline to Week 24
  This is a composite measure. Endpoints: SES-CD score, Robarts Histopathology Index score (measures histological disease activity; higher scores indicate more severe disease activity)
Comparison of the evolution of the faecal and mucosa-associated microbiota in participants with CD treated with EXL01 to participants treated with placebo (Part B only) | Maintenance Period Baseline to Week 24
  This is a composite measure. 16S sequencing / shotgun metagenomics and specific quantitative polymerase chain reaction (qPCR)/digital droplet (dd)PCR

CONTACTS AND LOCATIONS:
Overall Officials: Acting Chief Medical Officer, Study Director — Exeliom Biosciences
Locations (5):
- CHU de Liege, Liège, Belgium
- Poland (4):
  - Zespół Poradni Specjalistycznych REUMED, Lublin
  - Centrum Medyczne "Medyk" Sp. zo.o. Sp.K, Rzeszów
  - Endoskopia Sp. z o. o., Ul. B.Chrobrego 6/8, Sopot
  - PlanetMed Sp.z.o.o. Gastroenterology, Ul.Lubinowa 12/8, Wroclaw

IPD SHARING:
Plan to Share IPD: No